CLINICAL TRIAL: NCT05784298
Title: Acute Effect of Low-intensity Gamma Repetitive Transcranial Magnetic Stimulation on Cognitive and EEG Parameters in Older Adults With Mild Dementia by Alzheimer's Disease: a Randomized, Double-blind, Crossover, Controlled Trial
Brief Title: Acute Effect of Low-intensity Gamma rTMS on Cognitive and EEG Parameters in Adults With Mild Dementia by Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GER-4088-22-23-1
Record Dates: First submitted 2022-08-31; First posted 2023-03-24 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer Disease; Mild Dementia
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real low-intensity rTMS (Experimental): One 45 minutes session of stimulation. The stimulation coil will be located in the precuneus, located in the Pz area of the 10-20. The coil will emit a pulsed magnetic field at a frequency of 40 Hz with a magnetic field strength of 150 gauss.
  Interventions: Device: low-intensity rTMS
- Sham low-intensity rTMS (Sham Comparator): One 45 minutes session of stimulation. The stimulation coil will be located in the precuneus, located in the Pz area of the 10-20. The coil will not emit any magnetic field.
  Interventions: Device: low-intensity rTMS

INTERVENTIONS:
Device: low-intensity rTMS — 40 hz, 150 gauss, 1 session that lasts 45 minutes.

SUMMARY:
Neurocognitive disorders have a growing prevalence and impact on public health; their main etiology corresponds to Alzheimer's disease. To date, there is no treatment that can reverse neuronal damage in these pathologies. However, several non-invasive neuromodulation techniques, including transcranial magnetic stimulation, have been proposed as a viable option to halt the progression of the disease.

Transcranial magnetic stimulation (TMS) is a noninvasive, nonpainful neurostimulation technique with a high safety profile that has been successfully used to improve cognitive function in subjects with mild cognitive impairment. Our research group conducted a study that showed that the use of low-intensity TMS at gamma frequencies is a safe, non-invasive method with minimal adverse effects.

The present protocol proposes a new randomized, double-blind, crossover trial to be conducted in memory clinic patients over 65 years of age who meet the diagnosis of mild dementia due to Alzheimer's disease. The main objective is to evaluate the short-term cognitive and electroencephalographic changes produced by low-intensity, gamma-frequency transcranial magnetic stimulation.

A TMS device that emits a pulsed magnetic field at a frequency of 40 Hz, with a maximum magnitude of 150 gauss for 45 minutes will be used as an intervention. The intervention will be of two types, real or simulated, and will be applied twice to each patient, that is, in one session they will receive the real stimulation and in another the simulated one. In addition, during the sessions, cognitive and electroencephalographic measurements will be taken before, during and after each intervention. Each of these stimulation sessions should be separated by at least one week.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Age over 65 years old
* Who give written informed consent
* Patients with a diagnosis compatible with mild dementia according to NINCDS-ADRDA (National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association, 1984) criteria.
* CDR 1
* Preserved or corrected ability to see and hear
* Have a formal or informal caregiver

Exclusion Criteria:

* Clinical diagnosis of a neurodegenerative disease other than mild dementia due to Alzheimer's disease
* Present an uncontrolled medical condition at the time of the assessment for admission to the protocol (diabetes, heart disease, hypertension, hypothyroidism, uncontrolled renal or hepatic insufficiency).
* Diagnosis of major depression and/or some other untreated psychiatric illness (calculated with GDS)
* Excessive alcohol use
* Current or recent (6 months) use of any neurostimulation methods
* Metal implants excluding dental
* Signs or symptoms of increased intracranial pressure
* History of having received electroconvulsive therapy.
* Suffering from epilepsy.
* Having a deep brain stimulator implanted.
* Having any metallic prosthesis in the head.
* Having a pacemaker
* Extensive tattoos
* Taking any of the following medications:
* Tricyclic antidepressants such as: imipramine, amitriptyline, doxepin, nostriptyline, matroptyline.
* Antivirals such as: foscarnet, ganciclovir, ritonavir, dissociative anesthetics such as: phencyclidine, ketamine, γ-hydroxybutyrate
* Other stimulant drugs such as: amphetamines, cocaine, MDMA (ecstasy)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Changes in EEG gamma band activity | Baseline (1 second before stimulation burst) - Post (1 second after stimulation burst)

SECONDARY OUTCOMES:
Changes in Face-Name Associative Memory Test scores | Baseline (the last 10 minutes of the intervention) - Post (one week later, the last 10 minutes of the intervention)
  The Face-Name Associative Memory Test is a cross-modal associative memory test, it includes 20 face-name pairs. The administration procedure starts with the presentation of 20 faces with each name and participants should read the name underneath the faces and try to learn each face-name pair. After 5 minutes, the faces are shown one by one and participants are asked to recall the associated names from 4 different names. The correct number of pairs recalled is recorded.
Change from baseline in phonological and semantic verbal fluency test | Baseline (immediately before the intervention) - Post (Immediately after the intervention: 60 minutes approximately)
  The participant must say the largest number of words of a semantic category for one minute and then the largest number of words beginning with a given phoneme, also for one minute.
  Two versions of these tests are applied, one during baseline and one after stimulation.
  The order of application of the versions changes in the first and second sessions. That is, if in the first session they started with version 1 in the baseline and version 2 in the post, then in the second session they will start with version 2 and then version 1.
  There is a one week difference between the first and second session.
  The results obtained in the stimulation session and the sham session will be compared.
Changes in Rey Auditory Verbal Learning Test scores | Baseline (immediately before the intervention) - Post (Immediately after the intervention: 60 minutes approximately))
  Participants are given a list of 15 unrelated words repeated over five different trials and are asked to repeat. Another list of 15 unrelated words are given and the patient must again repeat the original list of 15 words and then again after 20 minutes.
  The score ranges from 0 (worse performance) to 15 (best performance).
  Two versions of this test are applied, one during baseline and one after stimulation.
  The order of application of the versions changes in the first and second sessions. That is, if in the first session one started with version 1 at baseline and version 2 at post, in the second session one will start with version 2 and then version 1.
  There is a one week difference between the first and second session.
  The results obtained in the stimulation session and the sham session will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mimenza-Alvarado AJ, Aguilar-Navarro SG, Abarca-Jimenez IE, Vazquez-Villasenor I, Luna-Umanzor DI, Dorard C, Villafuerte G. Low intensity gamma-frequency TMS safely modulates gamma oscillations in probable mild Alzheimer's dementia: a randomized 2 x 2 crossover pilot study. Front Neurol. 2025 May 15;16:1566476. doi: 10.3389/fneur.2025.1566476. eCollection 2025. PMID 40443505